CLINICAL TRIAL: NCT04835701
Title: Music as a Nonpharmacologic Approach to Pain Control With Intrauterine Device Placement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited staffing support to continue screening and enrollment process
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Melissa Lozano, Assistant Professor, Obstetrics, Gynecology and Reproductive Science, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-20-03749
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Contraception
Keywords: Intrauterine device; IUD; Pain; Music
MeSH Terms: conditions — Pain | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Intervention group (Experimental): Subjects randomized to the music group will choose 10 songs, which will be played during the procedure, from the time of positioning through completion of IUD insertion and speculum removal. Participants will otherwise undergo standard protocol for IUD insertion in an outpatient clinic setting. Total participation is predicted to last approximately 30 minutes.
  Interventions: Behavioral: Music
- Control group (No Intervention): Participants to undergo same standard protocol for IUD insertion in an outpatient clinic setting. No music will be played during the procedure.

INTERVENTIONS:
Behavioral: Music — Music may be played through a portable speaker in close proximity to the patient or through the patient's own headphones, if preferred. Music will be played at a low enough volume for subjects to hear standard anticipatory guidance during the procedure.
  Arms: Music Intervention group

SUMMARY:
The intervention of this study is the addition of patient-selected music during IUD insertion procedure. Subjects randomized to the music group will choose 10 songs, which will be played during the procedure, from the time of positioning through completion of IUD insertion and speculum removal. Music may be played through a portable speaker in close proximity to the patient or through the patient's own headphones, if preferred. Music will be played at a low enough volume for subjects to hear standard anticipatory guidance during the procedure. Both control and music groups will otherwise undergo the same standard protocol for IUD insertion in an outpatient clinic setting. Total participation is predicted to last approximately 30 minutes.

Subjects in both control and intervention groups will undergo the same assessment of pain during IUD insertion using the 100-mm visual analog scale (VAS). This will be administered at 8 points during the procedure. All subjects will also answer the same 5-question satisfaction survey following IUD insertion. Pain scores will be measured and compared between music and control groups to assess the primary and secondary outcomes of this study.

DETAILED DESCRIPTION:
This is a prospective, two-center, randomized controlled trial evaluating whether music reduces pain and improves satisfaction during IUD insertion. Computer-generated randomization assignments will allocate subjects to either music or standard protocol groups. 40 music and 40 control designations will be allocated to both sites, and all designations will be block-stratified into 10 blocks, each containing 4 controls and 4 intervention (music) subjects. This will ensure there are close to equal numbers of subjects in both groups if recruitment is halted before the minimum of 80 patients are enrolled. Assignments are available in a read-only document accessible by all co-investigators at the time of enrollment and randomization.

Subjects randomized to the music group will choose 10 songs, which will be played during the procedure, from the time of positioning through completion of IUD insertion and speculum removal. Music may be played through a portable speaker in close proximity to the patient or through the patient's own headphones, if preferred. Both control and music groups will otherwise undergo the same standard anticipatory guidance and protocol for IUD insertion in an outpatient clinic setting. Total participation is predicted to last approximately 30 minutes, as is standard for an appointment for IUD insertion. Study subjects will not interact with other participants.

Patients in both control and intervention groups will undergo intrauterine device (IUD) insertion. Pain will be assessed using a 100-mm visual analog scale (VAS) at 8 points during the procedure, including: (1) anticipated pain, (2) baseline pain prior to IUD insertion, (3) after speculum placement, (4) on tenaculum application, (5) on uterine sounding, (6) at IUD insertion, (7) after speculum removal, and (8) 5 minutes following the procedure. Patients will also answer a brief 5-question satisfaction survey following IUD insertion. Pain scores will be measured and compared between music and control groups to assess the primary and secondary outcomes of this study.

VAS scores will be recorded by the attending physician or co-investigator, as they will reliably note when each step of the procedure occurs and pain should be assessed. They will present the 100mm visual analog scale (VAS) to the patient at each of the 8 points of the procedure, and the patient will mark their pain score. Scores will be measured and documented by a single co-investigator to eliminate bias or differences in measurement.

VAS scores will be analyzed separately for each of the 8 distinct points described during the IUD insertion procedure. Differences between the intervention (music) and control groups will be assessed using a 0.05 level Wilcoxon ranksum test. A significant difference in pain will be noted if at least a 20 mm difference in VAS pain score exists between the two groups at any point of the procedure when VAS score is collected.

The aim of this study is to determine if music, chosen by the patient and played during IUD insertion, leads to lower pain scores and improved patient satisfaction with the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Nulliparous adult females age 18 years or older (nulliparous is defined as no prior pregnancies greater than or equal to 20 weeks of gestation)
* English-speaking patients
* Undergoing insertion of a copper or levonorgestrel intrauterine device
* Willing to comply with all study procedures

Exclusion Criteria:

* Non-English speaking patients
* Patients with a support person in the room during IUD insertion
* Patients desiring a paracervical block for analgesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 2. Nulliparous adult females age 18 years or older (nulliparous is defined as no prior pregnancies greater than or equal to 20 weeks of gestation)
Enrollment: 8 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
100-mm visual analog scale (VAS) | Day 1, at time of IUD insertion
  100-mm VAS total scale from 1-100 with higher score indicating more pain

SECONDARY OUTCOMES:
100-mm visual analog scale (VAS) | Day 1, baseline prior to IUD insertion
  100-mm VAS total scale from 1-100 with higher score indicating more pain
100-mm visual analog scale (VAS) | Day 1, after speculum placement
  100-mm VAS total scale from 1-100 with higher score indicating more pain
100-mm visual analog scale (VAS) | Day 1, on tenaculum application
  100-mm VAS total scale from 1-100 with higher score indicating more pain
100-mm visual analog scale (VAS) | Day 1, on uterine sounding
  100-mm VAS total scale from 1-100 with higher score indicating more pain
100-mm visual analog scale (VAS) | Day 1, after speculum removal
  100-mm VAS total scale from 1-100 with higher score indicating more pain
100-mm visual analog scale (VAS) | Day 1, 5 minutes following the procedure
  100-mm VAS total scale from 1-100 with higher score indicating more pain
Patient Satisfaction Survey | Day 1, post procedure at 30 minutes
  Patient Satisfaction Survey consists of 5-question administered post-procedure. Full scale from 1 to 5, with higher score indicating higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Neha R Bhardwaj, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Mount Sinai Beth Israel, New York, New York
  - Mount Sinai West, New York, New York

IPD SHARING:
Plan to Share IPD: No